CLINICAL TRIAL: NCT05493813
Title: Target-controlled Total Intravenous Anesthesia With Propofol Versus Sevoflurane Anesthesia for Endovascular Thrombectomy Procedure in Acute Ischemic Stroke Patients: Comparison of the Outcomes
Brief Title: Total Intravenous Anesthesia Versus Sevoflurane Anesthesia for Endovascular Thrombectomy in Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPEVGH IRB No.: 2021-04-001B
Record Dates: First submitted 2022-05-23; First posted 2022-08-09 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Ischemic Stroke, Acute; Thrombectomy; General Anesthesia; Total Intravenous Anesthesia; Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: ischemic stroke; general anesthesia; total intravenous anesthesia; postoperative delirium; postoperative cognitive dysfunction
MeSH Terms: conditions — Ischemic Stroke; Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-centered, double-blind, randomized control trial at Taipei Veterans General Hospital. Patients who are scheduled to undergo emergent EVT for acute ischemic stroke with large vessel occlusion will be randomly assigned to either of the two intra-procedural general anesthetic regimens that include a volatile anesthesia with sevoflurane (Sev-GA) or to a total intravenous anesthesia with propofol (TIVA-propofol).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients who meet the enrollment criteria and who provide written informed consent will be randomly assigned to either of the intubated Sev-GA or non-intubated TIVA-propofol groups according to either the discretion of anesthesiologist in charge or random allocation. If the patient was in critical situation, uncooperative, or with uncontrolled movement, the anesthesiologist would choose the intubated Sev-GA instead of the scheduled randomization. However, if patient is cooperative and not critical, the patient would be randomly assigned according to the randomization list created with the use of computer-generated, permuted-block sequences. Only the anesthesiologist and physicians involved in EVT are aware of the anesthesia assignment. On the contrary, patients, personnel who collect data, fill out questionnaire and scale measurement, and personnel who assess outcomes are unaware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubated Sevoflurane-GA group (Active Comparator): After preoxygenation for 3 minutes with 100% oxygen, anesthesia is induced with intravenous injection of propofol (1.5-2 mg/kg), remifentanil infusion (Ce value around 1-1.5 ng/kg), and cisatracurium (0.15-0.2 mg/kg), and followed by endotracheal intubation. General anesthesia is maintained with cisatracuirum (0.03 mg/kg every 45-50 min), remifentanil (Ce value around 1-1.5 ng/kg) and sevoflurane inhalation. Sevoflurane concentration will be adjusted to keep BIS value within the range of 40-60. Mechanical ventilation will be processed at volume-controlled mode with fraction of inspired oxygen (FiO2) 60%, tidal volume 6 ml/kg, and respiratory rate 9-12/min to keep normocapnia and avoid desaturation during the EVT procedure.
  Interventions: Behavioral: Cognitive function and delirium evaluation; Behavioral: Neurological functional assessment
- Non-intubated TIVA-propofol group (Active Comparator): With the application of Optiflow nasal high flow set at a flow rate of 20 L/min and 60% FiO2, total intravenous anesthesia is induced with target-controlled infusion of propofol (effect site (Ce) concentration around 1.5-2 μg/ml) and remifentanil (Ce value around 1.0-1.5 ng/ml), and adjusted as required.
  Interventions: Behavioral: Cognitive function and delirium evaluation; Behavioral: Neurological functional assessment

INTERVENTIONS:
Behavioral: Cognitive function and delirium evaluation — Cognitive functions (including delirium) will be assessed pre-procedure (baseline) and emergency department (before EVT), on day 1 and 7 and 3 months after EVT procedure
  Other Names: Confusion assessment method (CAM)
Behavioral: Neurological functional assessment — National Institute of Health Stroke Scale (NIHSS) and modified Rankin scale (mRS) will be assessed before (baseline but after stroke) and after EVT on days 1 and 7 after procedure up to 3 months follow-up.
  Other Names: National Institute of Health Stroke Scale (NIHSS) and modified Rankin scale (mRS)

SUMMARY:
The present clinical trial compares the effect of two general anesthesia (GA) modalities, the one with volatile anesthetic sevoflurane (endotracheal-intubated) and the other integrating total intravenous anesthesia (TIVA) with propofol (non-intubated), on post-procedural delirium and cognitive dysfunction after endovascular thrombectomy (EVT) in the participants with acute ischemic stroke. To assess the outcome of both modalities, the sedation depth of GA will be regulated with processed electroencephalogram monitor to reduce the incidence of postoperative delirium and the peri-procedural blood pressure will be controlled according to the guideline.Based on that, the investigators try to find a better general anesthetic modality for acute ischemic stroke participants undergoing EVT.

DETAILED DESCRIPTION:
1. In 2019, cerebrovascular disease (i.e., stroke) was the second leading cause of death worldwide.
2. The present guidelines for the early management of the participants with acute ischemic stroke urge the in-time and early application of intravenous chemical thrombolysis and endovascular thrombectomy (EVT) due to better outcome and prognosis. "Timing is brain."
3. The participants with acute ischemic stroke, previous stroke, and severe stroke have high incidence of delirium, and the stroke-related delirium has been shown to correlate with higher morbidity and mortality.
4. Researches on the anesthetic management during EVT for acute ischemic stroke have shown that both general anesthesia and sedation anesthesia are safe and without difference in neurological outcome and long-term complications. However, general anesthesia might have higher rates in revascularization in EVT for acute ischemic stroke as compared with sedation anesthesia.
5. Anesthesia could produce postoperative cognitive dysfunction (POCD) or delirium (POD), and general anesthesia could produce higher rates of POCD and POD compared to general anesthesia and sedation anesthesia. Additionally, brain injury and acute ischemic stroke are independent risk factors for POCD and POD. Whether the anesthetic management for EVT would interfere with the acute ischemic stroke-produced POCD and/or POD or even delay the detection and treatment of stroke-related neurological impairment deserves investigation since EVT is the gold standard for acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke with large vessel occlusion who are scheduled to undergo endovascular thrombectomy procedure, and
* Must be age of 20 to 90
* Must fulfill the indications for endovascular thrombectomy in acute ischemic stroke according to the American Heart Association/American Stroke Association 2018 Guidelines for the early management of patients with acute ischemic stroke and 2019 Taiwan stroke society guideline for endovascular thrombectomy in acute ischemic stroke, and
* Must agree to enroll into the clinical trial and sign the written informed consent from patients or delegates

Exclusion Criteria:

* Allergy to allergy to the anesthetics used in this clinical study
* Refusal for enrolling in study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive function and delirium evaluation | Baseline
  Cognitive functions (including delirium) will be assessed with the confusion assessment method. It is a validated delirium diagnostic tool, and is considered the "gold standard" for detection of delirium.: The four features of delirium are:1) acute onset and fluctuating course, 2) inattention, 3) disorganized thinking and 4) altered level of consciousness. A positive diagnosis of delirium is made if the person has feature 1 & 2 plus either 3 or 4. A positive diagnosis of delirium means that the patient's outcome is poor.
Change in Cognitive function and delirium evaluation | Day 1 after procedure
  Cognitive functions (including delirium) will be assessed with the confusion assessment method. It is a validated delirium diagnostic tool, and is considered the "gold standard" for detection of delirium.: The four features of delirium are:1) acute onset and fluctuating course, 2) inattention, 3) disorganized thinking and 4) altered level of consciousness. A positive diagnosis of delirium is made if the person has feature 1 & 2 plus either 3 or 4. A positive diagnosis of delirium means that the patient's outcome is poor.
Change in Cognitive function and delirium evaluation | Day 7 after procedure
  Cognitive functions (including delirium) will be assessed with the confusion assessment method. It is a validated delirium diagnostic tool, and is considered the "gold standard" for detection of delirium.: The four features of delirium are:1) acute onset and fluctuating course, 2) inattention, 3) disorganized thinking and 4) altered level of consciousness. A positive diagnosis of delirium is made if the person has feature 1 & 2 plus either 3 or 4. A positive diagnosis of delirium means that the patient's outcome is poor.
Change in Cognitive function and delirium evaluation | Month 3 after procedure
  Cognitive functions (including delirium) will be assessed with the confusion assessment method. It is a validated delirium diagnostic tool, and is considered the "gold standard" for detection of delirium.: The four features of delirium are:1) acute onset and fluctuating course, 2) inattention, 3) disorganized thinking and 4) altered level of consciousness. A positive diagnosis of delirium is made if the person has feature 1 & 2 plus either 3 or 4. A positive diagnosis of delirium means that the patient's outcome is poor.

SECONDARY OUTCOMES:
Neurological function: National Institute of Health Stroke Scale | Baseline
  National Institute of Health Stroke Scale (NIHSS) is widely used as a clinical assessment tool to evaluate acuity of stroke patients, being a predictor of both short and long term outcome of stroke patients, determine appropriate treatment, and predict patient outcome. Scores range from 0 to 42, with higher scores indicating greater severity: score 1-5 as mild, 5-14 as mild to moderately severe, 15-24 as severe, and > 25 as very severe situation.
Neurological function: National Institute of Health Stroke Scale | Day 1 after procedure
  National Institute of Health Stroke Scale (NIHSS) is widely used as a clinical assessment tool to evaluate acuity of stroke patients, being a predictor of both short and long term outcome of stroke patients, determine appropriate treatment, and predict patient outcome. Scores range from 0 to 42, with higher scores indicating greater severity: score 1-5 as mild, 5-14 as mild to moderately severe, 15-24 as severe, and > 25 as very severe situation.
Neurological function: National Institute of Health Stroke Scale | Day 7 after procedure
  National Institute of Health Stroke Scale (NIHSS) is widely used as a clinical assessment tool to evaluate acuity of stroke patients, being a predictor of both short and long term outcome of stroke patients, determine appropriate treatment, and predict patient outcome. Scores range from 0 to 42, with higher scores indicating greater severity: score 1-5 as mild, 5-14 as mild to moderately severe, 15-24 as severe, and > 25 as very severe situation.
Neurological function: National Institute of Health Stroke Scale | Month 3 after procedure
  National Institute of Health Stroke Scale (NIHSS) is widely used as a clinical assessment tool to evaluate acuity of stroke patients, being a predictor of both short and long term outcome of stroke patients, determine appropriate treatment, and predict patient outcome. Scores range from 0 to 42, with higher scores indicating greater severity: score 1-5 as mild, 5-14 as mild to moderately severe, 15-24 as severe, and > 25 as very severe situation.
Neurological function: modified Rankin scale | Baseline
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scores range from 0 to 6, with higher scores indicating greater severity:
  0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Neurological function: modified Rankin scale | Day 1 after procedure
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scores range from 0 to 6, with higher scores indicating greater severity:
  0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Neurological function: modified Rankin scale | Day 7 after procedure
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scores range from 0 to 6, with higher scores indicating greater severity:
  0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Neurological function: modified Rankin scale | Month 3 after procedure
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scores range from 0 to 6, with higher scores indicating greater severity:
  0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead

CONTACTS AND LOCATIONS:
Overall Officials: Hsu Ma, MD, PhD, Study Chair — Institutional Review Board, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No